CLINICAL TRIAL: NCT01911442
Title: A 6-Week, Randomized, Parallel, Double-Blind, Placebo-Controlled, Fixed-Dose, Multicenter Study to Evaluate the Efficacy and Safety of Lurasidone in Children and Adolescent Subjects With Irritability Associated With Autistic Disorder
Brief Title: Lurasidone Pediatric Autism Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D1050325
Record Dates: First submitted 2013-07-22; First posted 2013-07-30 (Estimated); Results first posted 2016-02-25 (Estimated); Last update posted 2016-02-25 (Estimated); Status verified 2016-01

CONDITIONS: Autism
Keywords: Autism, Lurasidone, Latuda
MeSH Terms: conditions — Autistic Disorder | interventions — Lurasidone Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Lurasidone 20 mg (Experimental): Lurasidone 20 mg once daily
  Interventions: Drug: Lurasidone 20 mg daily
- Lurasidone 60 mg (Experimental): Lurasidone 60 mg once daily
  Interventions: Drug: Lurasidone
- Placebo (Placebo Comparator): Placebo once daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lurasidone 20 mg daily — Lurasidone 20 mg once daily
  Other Names: Latuda
  Arms: Lurasidone 20 mg
Drug: Lurasidone — Lurasidone 60 mg once daily
  Other Names: Latuda
  Arms: Lurasidone 60 mg
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled study designed to evaluate the efficacy and safety of 2 fixed doses of lurasidone (20 mg/day and 60 mg/day) for 6 weeks compared with placebo in pediatric and adolescent subjects with irritability associated with autistic disorder who reside in the community setting.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled study designed to evaluate the efficacy and safety of 2 fixed doses of lurasidone (20 mg/day and 60 mg/day) for 6 weeks compared with placebo in pediatric and adolescent subjects with irritability associated with autistic disorder who reside in the community setting.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent from parent(s) or legal guardian(s) with sufficient intellectual capacity to understand the study and support subjects' adherence to the study procedures must be obtained for subjects who are not emancipated. In accordance with Institutional Review Board (IRB) requirements, the subject will complete an informed assent when developmentally appropriate, to participate in the study before conduct of any study-specific procedures.
* Male or female subjects 6 to 17 years of age, inclusive, at the time of consent.
* A reliable informant (eg, parent, legal guardian, or caregiver) who has past and current direct knowledge of the subject must accompany the subject at each visit and must oversee the administration of the study drug.
* DSM-IV-TR primary diagnosis of autistic disorder confirmation of the diagnosis by a trained clinician (eg, psychiatrist, psychologist, social workers, etc) at the time of screening, by means of the Autism Diagnostic Interview, Revised (ADI-R).
* Screening and Baseline ABC irritability subscale score ≥ 18.
* Screening and Baseline CGI-S ≥ 4.
* Within 5th to 95th percentile for gender specific Growth Charts from Centers for Disease Control (CDC).
* No clinically relevant abnormal laboratory values.
* No clinically relevant abnormal vital sign values/findings

  1. Females who participate in this study:

     * are unable to become pregnant (eg, premenarchal, surgically sterile, etc.) -OR-
     * practices true abstinence (consistent with lifestyle) and must agree to remain abstinent from signing informed consent to at least 7 days after the last dose of study drug has been taken;

-OR-

•are sexually active and willing to use a medically effective method of birth control (eg, male using condom and female using condom, diaphragm, contraceptive sponge, spermicide, contraceptive pill, or intrauterine device) from signing informed consent to at least 7 days after the last dose of study drug has been taken.

* Males must be willing to remain sexually abstinent (consistent with lifestyle) or use an effective method of birth control (eg, male using condom and female using condom, diaphragm, contraceptive sponge, spermicide, contraceptive pill, or intrauterine device) from signing informed consent to at least 7 days after the last dose of study drug has been taken.
* In the judgment of the investigator, the subject is able to swallow the size and number of study drug tablets specified per protocol (See Table 4 for study drug tablet size).
* Able to adhere to protocol-specified meal requirements during dosing.
* Have a stable living arrangement for at least 3 months prior to screening.
* Non-pharmacologic therapy (eg, behavior modification) must be stable for at least 4 weeks before screening and consistent throughout the study.

Exclusion Criteria:

* Subjects with profound intellectual disability.
* Current diagnosis of bipolar disorder, psychosis, schizophrenia or major depression, or childhood disintegrative disorder as confirmed by the MINI-Kid (as appropriate) at screening. Confirmed genetic disorders with cognitive and behavioral disturbances are also exclusionary.
* Clinically significant neurological, metabolic (including type 1 and type 2 diabetes), hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, carcinoma, and/or urological disorder that would pose a risk to the subjects if they were to participate in the study or that might confound the results of the study.

Note: Active medical conditions that are minor or well-controlled are not exclusionary if they do not affect risk to the subject or the study results. In cases in which the impact of the condition upon risk to the subject or study results is unclear, the Medical Monitor should be consulted. Any subject with a known cardiovascular disease or condition (even if controlled) must be discussed with the Medical Monitor during screening.

* Evidence of any chronic organic disease of the CNS such as tumors, inflammation, active seizure disorder, vascular disorder, potential CNS related disorders that might occur in childhood- eg, Duchenne Muscular dystrophy, myasthenia gravis, or other neurologic or serious neuromuscular disorders. In addition, subjects must not have a history of persistent neurological symptoms attributable to serious head injury. Past history of febrile seizure, drug-induced seizure, or alcohol withdrawal seizure is not exclusionary.
* If the subject has a history of seizures, the subjects must not currently be taking any antiepileptic drugs (AEDs) and be seizure-free for at least 6 months.
* Clinically significant finding(s) on physical examination determined by the investigator to pose a health concern to the subject while on study.
* A history or presence of abnormal ECG, which in the investigator's opinion is clinically significant. Screening ECGs will be centrally over-read, and eligibility will be determined based on the over-read.
* Known history or presence of clinically significant intolerance to any antipsychotic medications including but not limited to angioedema, serotonin or neuroleptic malignant syndromes, severe dystonia, or moderate to severe tardive dyskinesia.
* Clinically significant alcohol abuse/dependence or drug abuse/dependence based on Mini International Neuropsychiatric Interview for children and adolescents (MINI-Kid) criteria within the last 6 months prior to screening.
* Clinically significant orthostatic hypotension (ie, a drop in systolic blood pressure of 20 mmHg or more and/or drop in diastolic blood pressure of 10 mmHg or more within 4 minutes of standing up).
* Presence or history (within the last year) of a medical or surgical condition (eg, gastrointestinal disease) that might interfere with the absorption, metabolism, or excretion of orally administered lurasidone.
* Positive test results at screening for:

  1. Urine drugs of abuse (amphetamines, barbiturates, benzodiazepines, cocaine, opiates, phencyclidine, cannabinoids, methamphetamine, and methadone). However, a positive test for amphetamines, barbiturates, opiates, benzodiazepines or methadone may not result in exclusion of subjects if the investigator determines that the positive test is as a result of prescription medicine(s).
  2. Pregnancy test (only in female subjects ≥ 11 years old).
* Lifetime history of human immunodeficiency virus (HIV) positive or acquired immune deficiency syndrome (AIDS), or history of Hepatitis B or C.
* Participated in another interventional clinical trial or receiving an investigational product within 30 days prior to study drug administration.
* Use of concomitant medications that consistently prolong the QT/QTc interval within 28 days prior to randomization.
* Received depot neuroleptics unless the last injection was at least 1 month or 1 treatment cycle prior to screening, whichever is longer.
* Subject has received treatment with antidepressants within 3 days, fluoxetine hydrochloride at any time within 21 days, an MAO inhibitor within 21 days of randomization or clozapine within 120 days of randomization. Depot neuroleptics must be discontinued at least one treatment cycle prior to randomization.
* Use of any antipsychotic medication (other than study drug), carbamazepine, oxcarbazepine or fluvoxamine, within 3 days prior to randomization.
* Females who are pregnant, lactating, or likely to become pregnant during the study.
* Donation of whole blood within 60 days prior to randomization.
* Has a prolactin concentration greater than or equal to 100 ng/mL at screening.
* Subject is considered by the investigator to be at imminent risk of suicide during the study. Subject has a history of one or more serious suicide attempts (based on the investigator's judgment) in the 12 months prior to screening. Subjects determined to be at risk of suicide or injury, as assessed by the investigator at screening, will be referred for further psychiatric evaluation.
* Clinically relevant history of drug hypersensitivity to lurasidone or any components in the formulation.
* Subject requires use of concomitant medications that are potent inducers or inhibitors of the cytochrome P450 (CYP) 3A4 enzyme system (Appendix C) from signing informed consent until follow-up.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Actual)
Dates: Start 2013-08; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lurasidone Medical Director, MD, Study Director — Sumitomo Pharma America, Inc.
Locations (41):
- United States (41):
  - Harmonex Neuroscience Research, Dothan, Alabama
  - Southwest Autism Research & Resource Center, Phoenix, Arizona
  - Newport Beach Clinical Research Associates, Newport Beach, California
  - University of California San Francisco Medical Center, San Francisco, California
  - Florida Clinical Research Center, LLC, Bradenton, Florida
  - Sarkis Clinical Trials - Parent, Gainesville, Florida
  - Palm Springs Research Institute Inc, Hialeah, Florida
  - Florida Clinical Research Center, LLC, Maitland, Florida
  - Clinical Neuroscience Solutions, Inc., Orlando, Florida
  - Medical Research Group of Central Florida, Sanford, Florida
  - University of South Florida, St. Petersburg, Florida
  - University of South Florida, Tampa, Florida
  - Institute for Behavioral Medicine, LLC, Smyrna, Georgia
  - Capstone Clinical Research, Inc., Libertyville, Illinois
  - Baber Research Group, Naperville, Illinois
  - University of Kentucky, Lexington, Kentucky
  - Lake Charles Clinical Trials, LLC, Lake Charles, Louisiana
  - Kennedy Krieger Institute, Baltimore, Maryland
  - NeuroScientific Insights, Rockville, Maryland
  - Neurobehaviorial Medicine Group, PLLC, Bloomfield Hills, Michigan
  - Center for Psychiatry and Behavioral Medicine, Inc., Las Vegas, Nevada
  - Jersey Shore University Medical Center, Neptune City, New Jersey
  - Childrens Specialized Hospital, Toms River, New Jersey
  - Finger Lakes Clinical Research, Rochester, New York
  - Richmond Behavioral Associates, Staten Island, New York
  - Montefiore Medical Center PRIME, The Bronx, New York
  - Chapel Hill Neurology, Chapel Hill, North Carolina
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - The Ohio State University Nisonger Center, Columbus, Ohio
  - Cutting Edge Research Group, Oklahoma City, Oklahoma
  - Cyn3rgy Research & Development, Gresham, Oregon
  - Suburban Research Associates, Media, Pennsylvania
  - Segal Institute for Clinical Research, Charleston, South Carolina
  - Clinical Neuroscience Solutions, Inc., Memphis, Tennessee
  - Family Psychiatry of The Woodlands, P.A., The Woodlands, Texas
  - Ericksen Research & Development, LLC, Clinton, Utah
  - CRI Lifetree, Salt Lake City, Utah
  - University of Virginia, Charlottesville, Virginia
  - Neuroscience, Inc., Herndon, Virginia
  - Carilion Clinic, Roanake, Virginia
  - Pacific Institute of Medical Sciences, Bothell, Washington

REFERENCES:
- [Derived] Iffland M, Livingstone N, Jorgensen M, Hazell P, Gillies D. Pharmacological intervention for irritability, aggression, and self-injury in autism spectrum disorder (ASD). Cochrane Database Syst Rev. 2023 Oct 9;10(10):CD011769. doi: 10.1002/14651858.CD011769.pub2. PMID 37811711

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 46 centers in the United States between August 2013 and October 2014
Pre-assignment Details: Participants were screened and washed out up to 21 days.
Groups:
- Lurasidone 20 mg Once Daily: Subjects received 20 mg/day from Day 1 to Week 6 Visit
- Lurasidone 60 mg Once Daily: Subjects received lurasidone 20 mg/day from Days 1-3, 40 mg/day from Days 4-6 and 60 mg/day from Day 7 to Week 6 Visit. One-time dose reduction to Lurasidone 40 mg/day may occur in Weeks 2, 3 or 4 (ie, between Day 8 to Day 29, inclusive).
- Placebo: Subject received placebo to match lurasidone from Day 1 to Week 6 Visit
Period: Overall Study
Arm/Group | Lurasidone 20 mg Once Daily | Lurasidone 60 mg Once Daily | Placebo
Started | 49 | 51 | 50
Completed | 43 | 47 | 38
Not Completed | 6 | 4 | 12
Not completed — Adverse Event | 2 | 2 | 4
Not completed — Lack of Efficacy | 1 | 1 | 1
Not completed — Lost to Follow-up | 2 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 6
Not completed — Mother's Work Schedule | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The disposition table for the overall study used all subjects randomized. The baseline characteristics summary used safety population. 1 subject in placebo group did not take any study medication, and was removed from the safety population.
Groups:
- Lurasidone 20 mg Once Daily; Placebo: Subject received placebo to match lurasidone from Day 1 to Week 6 Visit
- Total: Total of all reporting groups
Arm/Group | Lurasidone 20 mg Once Daily | Lurasidone 60 mg Once Daily | Placebo | Total
Number analyzed (Participants) | 49 | 51 | 49 | 149
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 49 | 51 | 49 | 149
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 8 | 9 | 27
  Male | 39 | 43 | 40 | 122
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 7 | 7 | 25
  Not Hispanic or Latino | 38 | 44 | 42 | 124
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 0 | 2
  Asian | 0 | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 10 | 9 | 5 | 24
  White | 35 | 38 | 42 | 115
  More than one race | 0 | 1 | 1 | 2
  Unknown or Not Reported | 3 | 1 | 0 | 4
Region of Enrollment [Number; unit: participants]
  United States | 49 | 51 | 49 | 149

OUTCOME MEASURES:

1. Primary Outcome: Change in Aberrant Behavior Checklist (ABC) Irritability Subscale Score at Week 6
Description: The ABC irritability subscale score is the sum of 15 items, each rated among 0 = Not at all; 1 = Slight in degree; 2 = Moderately serious; and 3 = Severe in degree. The ABC irritability subscale score ranges from 0 to 45. Higher values of ABC subscale scores represent greater severity of illness.
Time Frame: Baseline to 6 Weeks
Population: Intent to treat (ITT) population includes all randomized subjects who receive at least one dose of study medication and have at least one post-baseline assessment in any efficacy variable.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Lurasidone 20 mg Once Daily | Lurasidone 60 mg Once Daily | Placebo
Number analyzed (Participants) | 48 | 51 | 49
units on a scale | 8.8 (1.5) | 9.4 (1.43) | 7.5 (1.52)
Statistical Analysis 1: Comparison: Lurasidone 20 mg Once Daily vs Placebo; LS Mean, LS mean difference and the associated 95% Cl and p-value for change from baseline are based on Mixed Model for Repeated Measures (MMRM); Test type: Superiority or Other; p = 0.5463, Mixed Models Analysis; Mean Difference (Final Values) = -1.3, 95% CI 2-sided [-5.6 to 3.0], Standard Error of Mean 2.15
Statistical Analysis 2: Comparison: Lurasidone 60 mg Once Daily vs Placebo; LS Mean, LS mean difference, and the associated 95% CI and p-value for change from baseline are based on Mixed Model for Repeated Measures; Test type: Superiority or Other; p = 0.3592, Mixed Models Analysis; Mean Difference (Final Values) = -1.9, 95% CI 2-sided [-6.1 to 2.2], Standard Error of Mean 2.09

2. Secondary Outcome: Change From Baseline in Clinical Global Impression-Severity (CGI-S) at Week 6
Description: The Clinical Global Impression - Severity of Illness (CGI-S) Scale is rated on a 7-point scale of severity with 1 = Normal, not at all ill to 7 = Among the most extremely ill patients. Higher values of CGI-S scores represent greater severity of illness.
Time Frame: Baseline to 6 Weeks
Population: Intent to treat population. 49 in the placebo arm is correct. One subject in the placebo group did not receive the study medication, and therefore that subject was removed from the ITT population. A total of 50 subjects were randomized and 49 subjects were included in the placebo group of the ITT population.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Lurasidone 20 mg Once Daily | Lurasidone 60 mg Once Daily | Placebo
Number analyzed (Participants) | 48 | 51 | 49
units on a scale | -1.1 (0.17) | -1.0 (0.16) | -0.7 (0.17)
Statistical Analysis 1: Comparison: Lurasidone 20 mg Once Daily vs Placebo; Test type: Superiority or Other; p = 0.1755, Mixed Models Analysis; Mean Difference (Final Values) = -0.3, Standard Error of Mean 0.25 — This is due to rounding. the LSM for Lurasidone 20 mg/d at week 6 was -1.069 vs -0.734 for placebo group. So the LSM of the treatment difference between Lurasidone 20 mg/d and placebo was 0.335 if 3 decimals are reported
Statistical Analysis 2: Comparison: Lurasidone 60 mg Once Daily vs Placebo; Test type: Superiority or Other; p = 0.2402, Mixed Models Analysis; Mean Difference (Final Values) = -0.3, Standard Error of Mean 0.24

3. Secondary Outcome: Change From Baseline in Aberrant Behavior Checklist (ABC) Hyperactivity Subscale Score at Week 6
Description: The ABC hyperactivity and noncompliance subscale score is the sum of 16 items, each rated among 0 = Not at all; 1 = Slight in degree; 2 = Moderately serious; and 3 = Severe in degree. The ABC hyperactivity and noncompliance subscale score may range from 0 to 48. In general, higher values of ABC subscale scores represent greater severity of illness.
Time Frame: Baseline to 6 Weeks
Population: ITT
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Lurasidone 20 mg Once Daily | Lurasidone 60 mg Once Daily | Placebo
Number analyzed (Participants) | 48 | 51 | 49
units on a scale | -9.7 (1.50) | -6.6 (1.43) | -7.1 (1.52)

4. Secondary Outcome: Change From Baseline in Children's Yale-Brown Obsessive Compulsive Scales (CY-BOCS) Modified for Pervasive Developmental Disorders (PDDs)
Description: CY-BOCS total score ranges from 0 to 20. The higher value of CY-BOCS scores the greater severity of illness. This table is a summary of Y-BOCS compulsion total score.
Time Frame: 6 Weeks
Population: ITT
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Lurasidone 20 mg Once Daily | Lurasidone 60 mg Once Daily | Placebo
Number analyzed (Participants) | 48 | 51 | 49
units on a scale | -1.0 (0.46) | -1.0 (0.44) | -1.2 (0.49)

5. Secondary Outcome: Change From Baseline in the Caregiver Strain Questionnaire (CGSQ)
Description: CGSQ is a caregiver reported assessment to assesses extent to which caregivers are affected by special demands associated with caring for a child with emotional/behavioral problems. CGSQ is comprised of three subscales which range in severity from 1 to 5 (Objective Strain, Subjective Externalized Strain, Subjective Internalized Strain), The 3 subscales are calculated as the averages of the corresponding individual items. Higher scores on each indicates greater strain. A Global Strain score is calculated by summing the three subscales (Objective Strain, Subjective Externalized Strain, Subjective Internalized Strain) to provide an indication of the total impact of the special demands on the family. Global Strain scores range from 3 to 15. As with the individual subscales, higher scores indicate greater strain.
Time Frame: 6 Weeks
Population: ITT
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Lurasidone 20 mg Once Daily | Lurasidone 60 mg Once Daily | Placebo
Number analyzed (Participants) | 48 | 51 | 49
units on a scale | -1.49 (0.292) | -1.66 (0.274) | -1.35 (0.300)

6. Secondary Outcome: Proportion of Subjects Who Have CGI-I Score of 1 (Very Much Improved) or 2 (Much Improved) at Week 6
Time Frame: 6 Weeks
Population: ITT - the current data presented is at week 6.
Measure: Number; unit: percentage of subjects
Arm/Group | Lurasidone 20 mg | Lurasidone 60 mg | Placebo
Number analyzed (Participants) | 43 | 47 | 38
percentage of subjects | 17 | 17 | 14

7. Secondary Outcome: Proportion of Subjects Who Have at Least 25% Reduction From Baseline to Week 6 in the ABC Irritability Subscale Score.
Time Frame: 6 Weeks
Population: ITT
Measure: Number; unit: percentage of subjects
Arm/Group | Lurasidone 20 mg | Lurasidone 60 mg | Placebo
Number analyzed (Participants) | 43 | 47 | 38
percentage of subjects | 25 | 26 | 23

ADVERSE EVENTS:
Time Frame: Adverse event data were collected as spontaneous reports at all visits
Description: Participant flow module presents all subjects randomized. The summary of AEs is based on safety population. As explained earlier, there were 49 placebo subjects included in the safety population.
Arm/Group | Lurasidone 20 mg Once Daily | Lurasidone 60 mg Once Daily | Placebo
Serious Adverse Events (participants affected / at risk) | 3/49 | 2/51 | 0/49
Other Adverse Events (participants affected / at risk) | 33/49 | 38/51 | 28/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lurasidone 20 mg Once Daily (N=49) | Lurasidone 60 mg Once Daily (N=51) | Placebo (N=49)
Torus Fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Upper Limb Fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Appendicitis (General disorders) | 0 (0) | 1 (1) | 0 (0)
Irritability (General disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lurasidone 20 mg Once Daily (N=49) | Lurasidone 60 mg Once Daily (N=51) | Placebo (N=49)
Vomiting (Gastrointestinal disorders) | 4 (4) | 14 (17) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 4 (4) | 4 (4)
Nausea (Gastrointestinal disorders) | 2 (2) | 3 (6) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 3 (3) | 1 (1)
Gastritis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Abdominal Discomfort (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 3 (4) | 9 (10) | 2 (2)
Akathisia (Nervous system disorders) | 3 (5) | 3 (6) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 3 (3) | 3 (4)
Psychomotor Hyperactivity (Nervous system disorders) | 2 (2) | 2 (2) | 1 (2)
Sedation (Nervous system disorders) | 3 (3) | 1 (1) | 1 (1)
Lethargy (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Disturbance in Attention (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Nasopharynigitis (Infections and infestations) | 5 (5) | 3 (4) | 0 (0)
Gastroenteritis Viral (Infections and infestations) | 1 (1) | 1 (1) | 2 (2)
Rhinitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Aggression (Psychiatric disorders) | 2 (3) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (1) | 5 (5)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3) | 2 (2)
Fatigue (General disorders) | 1 (1) | 4 (5) | 1 (1)
Pyrexia (General disorders) | 2 (2) | 1 (1) | 0 (0)
Irritability (General disorders) | 2 (2) | 0 (0) | 2 (2)
Laceration (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 1 (1)
Weight Increased (Investigations) | 1 (1) | 4 (4) | 1 (1)
Increased Appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 3 (3)
Enuresis (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
There IS agreement between Principal Investigator and Sponsor that restricts PI's rights to discuss or publish trial results after trial is completed.

In addition to the <60-180 day restriction above, since this is a multicenter study, 1st publication of study results shall be made with other participating study sites as a multicenter publication provided, if a multicenter publication is not forthcoming within 24 months post completion of study at all sites, PI shall be free to publish.